CLINICAL TRIAL: NCT05364944
Title: A Phase 1b Study in Patients With Acromegaly or Functioning Gastroenteropancreatic Neuroendocrine Tumors (GEP-NETs) to Characterize the Pharmacokinetics, Pharmacodynamics, Safety and Tolerability of Debio 4126, a 12-week Prolonged-release Octreotide Formulation
Brief Title: A Study to Assess the Pharmacokinetics, Pharmacodynamics, Safety, and Tolerability of Debio 4126 in Participants With Acromegaly or Functioning Gastroenteropancreatic Neuroendocrine Tumors (GEP-NETs)
Acronym: OXTEND-01
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The recruitment was halted for strategic reasons
Sponsor: Debiopharm International SA (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Debio 4126-102; 2021-005035-23 (EudraCT Number)
Record Dates: First submitted 2022-05-04; First posted 2022-05-06 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Acromegaly; GEP-NET
MeSH Terms: conditions — Acromegaly; Gastro-enteropancreatic neuroendocrine tumor | interventions — Octreotide; lanreotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort A: Participants With Acromegaly (Experimental): Participants will receive Sandostatin Long-acting repeatable (LAR) or Somatuline Autogel (ATG) (or equivalent formulations of octreotide/lanreotide) in Run-in Period and further will receive Debio 4126 in this group.
  Interventions: Drug: Debio 4126; Drug: Sandostatin LAR; Drug: Somatuline ATG
- Cohort B: Participants With GEP-NET (Experimental): Participants will receive Sandostatin LAR or Somatuline ATG (or equivalent formulations of octreotide/lanreotide) in Run-in Period and further will receive Debio 4126 in this group.
  Interventions: Drug: Debio 4126; Drug: Sandostatin LAR; Drug: Somatuline ATG

INTERVENTIONS:
Drug: Debio 4126 — Intramuscular (IM) injection
Drug: Sandostatin LAR — Sandostatin LAR will be administered as IM injection as pre-study treatment dose prior to Debio 4126 administration
  Other Names: Octreotide acetate
Drug: Somatuline ATG — Somatulin ATG will be administered as deep subcutaneous (SC) injection as pre-study treatment dose prior to Debio 4126 administration
  Other Names: Lanreotide acetate

SUMMARY:
This is an open-label, single treatment arm, multicenter study to assess the pharmacokinetics (PK), pharmacodynamics (PD), safety, and tolerability of Debio 4126 in the treatment of participants with Acromegaly or Functioning Gastroenteropancreatic Neuroendocrine tumors (GEP-NETs).

ELIGIBILITY:
Main Inclusion Criteria:

For Participants with Acromegaly:

* Treatment with octreotide LAR (≤30 mg dose once in 4 weeks [Q4W] IM) or lanreotide ATG (≤120 mg Q4W or 120 mg once in 6 weeks [Q6W] to once in 8 weeks [Q8W] as deep SC injection) for at least 6 months overall, and for at least 2 months at a stable dose as monotherapy for acromegaly treatment prior to entering Run-in (Day -28). Octreotide doses of 10, 20, and 30 mg are considered similar to lanreotide doses of 60, 90, and 120 mg. Thus, a switch between similar doses of the two products will be considered as the patient remaining on a stable dose, unless due to efficacy or safety
* Diagnosis of acromegaly by historical evidence of (persistent or recurrent) acromegaly will be carried out
* IGF-1 ≤1.3 x upper limit of normal (ULN) assessed centrally at screening

For Participants with GEP-NETs:

* Treatment with octreotide LAR (≤ 30 mg dose Q4W IM) or lanreotide ATG (≤ 120 mg Q4W or 120 mg Q6W to Q8W as deep SC injection) for at least 6 months overall, and for at least 2 months at a stable dose as monotherapy for study disease treatment prior to entering Run-in (Day -28). Octreotide doses of 10, 20, and 30 mg are considered similar to lanreotide doses of 60, 90, and 120 mg. Thus, a switch between similar doses of the two products will be considered as the participant remaining on a stable dose, unless due to efficacy or safety
* Participants with functioning, well-differentiated (Grade 1 or Grade 2) GEP-NET with symptoms of carcinoid syndrome which are controlled by Sandostatin LAR, Somatuline ATG, or equivalent medications; sporadic use of rescue medication for symptom control, e.g., bowel movements and/or flushing, is allowed

Main Exclusion Criteria:

For Participants with Acromegaly and GEP-NETs:

* Known ongoing gallbladder or bile duct disease or acute or chronic pancreatitis
* Hypothyroidism not adequately treated with thyroid hormone replacement therapy
* Diabetic participants whose blood glucose is poorly controlled despite adequate therapy, as evidenced by glycated hemoglobin (HbA1c) >8.0% at screening
* Cardiology:

  1. Known left ventricular ejection fraction <50%, left ventricular hypertrophy, ventricular arrhythmias, bradycardia (heart rate <50 beats per minute [bpm]), cardiomyopathy
  2. New York Heart Association Class ≥3 heart failure
  3. Congenital long QT syndrome or
  4. Known family history of long QT syndrome or sudden cardiac death before the age of 50
  5. Symptomatic Pulmonary embolism
  6. QT interval corrected for heart rate according to Fridericia's formula (QTcF) at screening >450 milliseconds (msec) for males and >470 msec for females, based on the average of a triplicate ECG

For Participants with Acromegaly:

* Participants who received pituitary irradiation <2 years prior to enrollment as stereotactic radiotherapy or <3 years prior to enrollment for conventional radiotherapy
* Participants who received medical treatment with pasireotide (within 6 months prior to screening), pegvisomant (within 3 months prior to screening), dopamine agonists (within 3 months prior to screening)
* Participants who have undergone pituitary surgery within 6 months prior to screening

For Participants with GEP-NETs:

* Participants with short-bowel syndrome
* Participants with poorly differentiated neuroendocrine carcinoma and/or high-grade neuroendocrine carcinoma
* Participants who have received any previous therapy with interferons, targeted therapies (e.g., everolimus, sunitinib, bevacizumab), chemotherapy or other anti-neoplastic systemic therapies administered for more than 1 month and within 12 weeks prior to the start of the Run-in period
* Participants having history of hepatic embolization, hepatic arterial chemoembolization, and/or selective internal radiation (SIR) therapy within less than 6 months prior to screening
* Participants who have received Peptide receptor radionuclide therapy (PRRT) therapy during the last 12 months prior to screening

[Note: Other inclusion/exclusion criteria mentioned in the protocol may apply.]

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2022-05-18 (Actual); Primary Completion 2024-10-29 (Actual); Study Completion 2024-12-03 (Actual)

PRIMARY OUTCOMES:
Plasma Concentration of Debio 4126 in Acromegaly and GEP-NET Participants | Predose at Days -28 to -7; Postdose at multiple timepoints from Day 1 to Day 337
  The PK of Debio 4126 will be evaluated in plasma.

SECONDARY OUTCOMES:
Assessment of Ratio of Accumulation (Rac) of Octreotide in Plasma After Repeated Administration of Debio 4126 in Acromegaly and GEP-NET Participants | Predose at Days -28 to -7; Postdose at multiple timepoints from Day 1 to Day 337
Safety and Tolerability of Debio 4126 as Assessed by Number of Participants With At Least one Treatment Emergent Adverse Events (TEAE) in Acromegaly and GEP-NET Participants | Up to Week 65
Local Tolerability of Debio 4126 as Assessed by Pain at Injection Site Based on Pain Visual Analog Scale (VAS) Score in Acromegaly and GEP-NET Participants | Up to Week 65
  Pain VAS scale score will be assessed on 4-point rating scale, where 0=absent and 3=severe.
Insulin-Like Growth Factor 1 (IGF-1) and Growth Hormone (GH) Levels in Acromegaly Participants | Baseline up to Week 48
  The blood samples will be collected to assess changes in the levels of IGF-1 (in µg/L) and GH (in µg/L).
Number of Participants With Carcinoid Syndrome Symptoms and use of Rescue Medication for Symptom Control in GEP-NET Participants | Baseline up to Week 48

CONTACTS AND LOCATIONS:
Locations (14):
- Rigshospitalet, Endokrinologisk afdeling, Copenhagen, Denmark
- France (3):
  - CHU Angers, Angers
  - AP-HP Hopital Bicetre, Le Kremlin-Bicêtre
  - AP-HM - Hôpital de la Conception, Service d'Endocrinologie et Centre de Référence des Maladies Rares de l'hypophyse, Marseille
- Medicover Praxis fur Neuroendokrinologie, Munich, Germany
- Israel (2):
  - Rabin Medical Center, Beilinson Hospital, Clalit Health Services by Rabin Medical Center, Beilinson Hospita, Petah Tikva
  - Sheba Medical Center, Endocrine institute, Ramat Gan
- Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico di Milano, Milan, Italy
- Poland (2):
  - Uniwersyteckie Centrum Kliniczne im. Prof. K. Gibinskiego Slaskiego Uniwersytetu Medycznego w Katowicach, Katowice
  - Mazowiecki Szpital Brodnowski - Zespol Oddzialow Chorob Wewnetrznych, Endokrynologii i Diabetologii, Warsaw
- Spain (2):
  - Hospital de la Santa Creu i Sant Pau Barcelon, Barcelona
  - Hospital Universitario Virgen del Rocio, Seville
- United Kingdom (2):
  - University Hospital Coventry, WISDEM Centre, UHCW NHS Trust, Coventry
  - Royal Free London NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: No